CLINICAL TRIAL: NCT02235337
Title: The Impact of Riboflavin on the Severity and Duration of Sports Related Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: James Madison University (Other)
Responsible Party: Principal Investigator, Jeremy Kent, MD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17406
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Sports Related Concussion
Keywords: Concussion; Sports related concussion; mTBI; Vitamin B; Riboflavin
MeSH Terms: conditions — Brain Concussion | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Riboflavin (Experimental)
  Interventions: Drug: Riboflavin 400mg daily

INTERVENTIONS:
Drug: Riboflavin 400mg daily
  Other Names: Vitamin B2

SUMMARY:
The purpose of this study is to investigate the effectiveness of riboflavin to decrease the duration of time for a student-athlete to return to participation in sports after a sports related concussion.

ELIGIBILITY:
Inclusion Criteria:

* All UVa and JMU student-athletes over the age of 18 years old who are diagnosed with a sports related concussion

Exclusion Criteria:

* Less than 18 years old
* Greater than 24 hours have elapsed since the concussion occurred.
* The student-athlete has already participated in the study during which he/she took Riboflavin
* Non-sports related concussion not incurred while participating in the sport or training for the sport. As an example, a student-athlete who sustains a concussion as a result of a motor vehicle accident will be excluded from the study for that concussion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Time to return to full participation in sports after a sports related concussion | 21 days or less

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Virginia, Charlottesville, Virginia
  - James Madison University, Harrisonburg, Virginia

REFERENCES:
- [Background] Barbre AB, Hoane MR. Magnesium and riboflavin combination therapy following cortical contusion injury in the rat. Brain Res Bull. 2006 May 31;69(6):639-46. doi: 10.1016/j.brainresbull.2006.03.009. Epub 2006 Apr 3. PMID 16716831
- [Background] Kokiko ON, Hamm RJ. A review of pharmacological treatments used in experimental models of traumatic brain injury. Brain Inj. 2007 Mar;21(3):259-74. doi: 10.1080/02699050701209964. PMID 17453754
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] MacLennan SC, Wade FM, Forrest KM, Ratanayake PD, Fagan E, Antony J. High-dose riboflavin for migraine prophylaxis in children: a double-blind, randomized, placebo-controlled trial. J Child Neurol. 2008 Nov;23(11):1300-4. doi: 10.1177/0883073808318053. PMID 18984840
- [Background] Maizels M, Blumenfeld A, Burchette R. A combination of riboflavin, magnesium, and feverfew for migraine prophylaxis: a randomized trial. Headache. 2004 Oct;44(9):885-90. doi: 10.1111/j.1526-4610.2004.04170.x. PMID 15447697
- [Background] McCrory P, Meeuwisse W, Aubry M, Cantu B, Dvorak J, Echemendia R, Engebretsen L, Johnston K, Kutcher J, Raftery M, Sills A, Benson B, Davis G, Ellenbogen R, Guskiewicz K, Herring SA, Iverson G, Jordan B, Kissick J, McCrea M, McIntosh A, Maddocks D, Makdissi M, Purcell L, Putukian M, Schneider K, Tator C, Turner M. Consensus statement on Concussion in Sport--the 4th International Conference on Concussion in Sport held in Zurich, November 2012. J Sci Med Sport. 2013 May;16(3):178-89. doi: 10.1016/j.jsams.2013.02.009. Epub 2013 Mar 29. No abstract available. PMID 23541595
- [Background] Patterson ZR, Holahan MR. Understanding the neuroinflammatory response following concussion to develop treatment strategies. Front Cell Neurosci. 2012 Dec 12;6:58. doi: 10.3389/fncel.2012.00058. eCollection 2012. PMID 23248582
- [Background] Schoenen J, Jacquy J, Lenaerts M. Effectiveness of high-dose riboflavin in migraine prophylaxis. A randomized controlled trial. Neurology. 1998 Feb;50(2):466-70. doi: 10.1212/wnl.50.2.466. PMID 9484373
- [Background] Sundaram U. Regulation of intestinal vitamin B(2) absorption. Focus on "Riboflavin uptake by human-derived colonic epithelial NCM460 cells". Am J Physiol Cell Physiol. 2000 Feb;278(2):C268-9. doi: 10.1152/ajpcell.2000.278.2.C268. No abstract available. PMID 10666021
- [Background] Trojian TH, Jackson E. Omega-3 polyunsaturated fatty acids and concussions: treatment or not? Curr Sports Med Rep. 2011 Jul;10(4):180-5. doi: 10.1249/JSR.0b013e31822458d5. No abstract available. PMID 23531891
- [Background] Yee AJ. Effectiveness of high-dose riboflavin in migraine prophylaxis. Neurology. 1999 Jan 15;52(2):431-2. doi: 10.1212/wnl.52.2.431-a. No abstract available. PMID 9932987